CLINICAL TRIAL: NCT02904044
Title: Etude Des Traumatismes Sportifs Lors Des Cours d'éducation Physique et Sportive Chez Les collégiens Dans le Sud de l'Ile de La Reunion
Brief Title: Sport Injuries During Physical Activity Lessons in Secondary School in South of Reunion Island
Acronym: TsColEPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/CHU/TsColEPS
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Athletic Injuries
Keywords: School; Sport; Injuries
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Injured/Case: Secondary school pupil injured during a physical activity lesson between 2012-2014 in south of Reunion Island
- Control: Same age and gender than case in the same classroom and during the same physical activity lesson

SUMMARY:
TsColEPS aims at identifying individual determinants of sport injuries during physical activity lessons in secondary school at reunion Island.

DETAILED DESCRIPTION:
Sport injuries during physical activities lessons are the first etiology of traumatism in secondary school. Epidemiological studies on individual determinants of sport injuries are very scarce and most focused on contextual or mixed determinants.

TsColEPS is a multicenter case control study with one control paired to one case.

A convenience sample of 500 pupils in each group was planned on the base of a range of expected odds ratios.

ELIGIBILITY:
Inclusion Criteria:

* in secondary public school classroom in south of Reunion Island
* no age limited

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Reunion Island secondary school pupils
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Individual determinants of sport injuries during physical activity lessons in secondary school measured by a series of questionnaires at school (nurse interview), at home (family interview) and at the doctor's office for diagnosis | 2 years with 1 year follow-up
  Questionnaires are compiled in the CRC for datamanagement and analysis. Determinants are computed in frequency and proportion or mean +/- SD and analysed in a multilevel model

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Saint-Pierre, Île de La Réunion, France

IPD SHARING:
Plan to Share IPD: Undecided